CLINICAL TRIAL: NCT07095270
Title: Evaluation of Circadian OS Technology on Melatonin Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Director, Light and Health Research Center at Mount Sinai, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-24-00822
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Circadian Disruption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Condition - iPad with Circadian OS App (Active Comparator): iPad with Circadian OS App ON - iPad screen brightness adjusted by Circadian OS software to provide circadian-effective light exposure.
  Interventions: Device: Circadian OS software
- Control Condition (Placebo Comparator): iPad with Circadian OS App OFF and iPad screen dimmed to lowest setting
  Interventions: Device: Circadian OS software

INTERVENTIONS:
Device: Circadian OS software — Circadian OS is a software program that runs on existing iPads. It utilizes the iPad capabilities to control and deliver circadian-effective light.

SUMMARY:
Primary Objective: Evaluate how the Circadian OS iPad-based light intervention suppresses melatonin. This small pilot study is designed to validate the Circadian OS technology by testing physiological response using melatonin suppression. The study aims to evaluate how the Circadian OS iPad-based light intervention influences sleepiness as measured objectively via suppression of melatonin and subjectively via the Karolinska Sleepiness scale.

DETAILED DESCRIPTION:
Aims: To test whether the Circadian OS app delivers sufficient circadian effective light that will result in measurable melatonin suppression (target suppression is 30% after 1 hour exposure)

Hypothesis: The Circadian OS app will deliver a Circadian Stimulus (CS) of 0.3 at the eye level and will result in 30% melatonin suppression after one hour using the device compared to less than 10% suppression without the Circadian OS app and the subjects will feel less sleepy (KSS score) when exposed to the Circadian OS app compared to no app

Outcomes: melatonin suppression will be calculated from saliva samples and subjective sleepiness as self-rated on the Karolinska Sleepiness Scale (KSS)

ELIGIBILITY:
Inclusion Criteria:

• Healthy adults over the age of 30

Exclusion Criteria:

* Use of over-the-counter melatonin or prescription medications
* Obstructing cataracts, macular degeneration, or blindness
* Heart disease or high blood pressure

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Melatonin Level | immediately prior to the iPad turning on, after 30 minutes of light exposure and after 60 minutes of light exposure
  Melatonin is a natural hormone that is mainly produced by a gland in the brain and helps regulate the body's natural sleep-wake cycle.

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale (KSS) | immediately prior to the iPad turning on, after 30 minutes of light exposure and after 60 minutes of light exposure
  Sleepiness using the Karolinska Sleepiness Scale (KSS) which includes one item - participants will rate how sleep they are feeling on a scale of 0 to 9,with higher score indicating being the most sleepy

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
no individual results will be shared, only overall averages